CLINICAL TRIAL: NCT00614757
Title: The Prevalence of Insulin Resistance and the Potential Modulation of Insulin Resistance by N-acetylcysteine (NAC) in Patients Chronically Infected by the Hepatitis C Virus
Brief Title: Insulin Resistance Study
Acronym: IR
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Biomedical Research Foundation (Other)
Responsible Party: Principal Investigator, Prashant Pandya, Principal Investigator, Kansas City Veteran Affairs Medical Center
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKP0003; 00173
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Insulin Resistance; Metabolic Syndrome x
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (No Intervention): One half of the patients will take not medication for 30 days and then have labs redrawn
- 1 (Experimental): one half of the patients with insulin resistance will take 4ml of 20% N-acetylcysteine BID for 30 days
  Interventions: Drug: N-acetylcysteine 20% 4ml; Drug: N-acetylcysteine 20% in 4 ml

INTERVENTIONS:
Drug: N-acetylcysteine 20% 4ml — N-acetylcysteine 20% 4ml
  Arms: 1
Drug: N-acetylcysteine 20% in 4 ml — N-acetylcysteine 20% in 4 ml
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate how often patients with hepatitis C infection have abnormalities of sugar and fat utilization. Additionally we would like to find out if these abnormalities of sugar and fat utilization are common in other liver diseases, or related to being overweight.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written consent
* HCV RNA PCR positive for 6 months
* Normal Hgb, WBC,Neutrophils
* Platelets of >/= 65,000
* Direct Bili, within 20% ULN
* Albumin >3
* Serum Creatinine <20% ULN
* TSH WNL
* AFP </= 100

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* No Thiazolidinedione, Metformin,unless required for the treatment of type II DM
* Hepatitis C of non-genotype 1,2,3
* Any other cause for liver disease other than chronic hepatitis C
* Hemoglobinopathies
* Evidence of advanced liver disease
* Previous organ transplant
* Severe psychiatric disorder
* Significant cardiovascular dysfunction within the past 12 months
* Poorly controlled diabetes mellitus
* Immunologically mediated disease
* Any medical condition requiring chronic systemic administration of steroids
* Evidence of an active or suspected cancer
* Substance abuse at the time of the study
* Known HIV
* Irritability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Those patients who are identified to have insulin resistance will be asked to participate in the treatment phase of the study | 2 years

SECONDARY OUTCOMES:
One half of patients with insulin resistance will undergo 30 day treatment with N-acetylcysteine to see if we can measure an improvement in fasting insulin and glucose levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Prashant K Pandya, DO, Principal Investigator — Kansas City VA Medical Center
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States